CLINICAL TRIAL: NCT00539955
Title: Brief Intervention to Reduce Drinking Among Batterers
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Tennessee, Knoxville (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Butler Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIAAA-STU_014193_0111-001-M; R01AA014193 (NIH)
Record Dates: First submitted 2007-09-25; First posted 2007-10-05 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Intimate Partner Violence; Alcohol Use
Keywords: intimate partner violence; alcohol use; substance use
MeSH Terms: conditions — Alcohol Drinking; Substance-Related Disorders | interventions — Ethanol; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Other): Standard 40 hour state-mandated batterer intervention
  Interventions: Behavioral: Standard Batterer Intervention
- 2 (Other): Brief alcohol intervention combined with standard batterer intervention
  Interventions: Behavioral: Brief Alcohol Intervention

INTERVENTIONS:
Behavioral: Standard Batterer Intervention — Standard state-mandated batterer intervention program (40 hours)
  Arms: 1
Behavioral: Brief Alcohol Intervention — Brief alcohol intervention combined with state mandated batterer intervention program
  Arms: 2

SUMMARY:
The goal of this project is to examine whether, relative to standard care, violence and alcohol use outcomes can be improved by a brief, motivationally based adjunct alcohol treatment for men enrolled in batterer intervention programs. We hypothesize that men randomized to also receive the brief alcohol intervention will have better partner violence and alcohol use outcomes than men who are randomized to the batterer intervention program alone.

ELIGIBILITY:
Inclusion Criteria:

* Participation in a batterer intervention program
* Hazardous drinking

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 253 (Estimated)
Dates: Start 2003-07; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Intimate partner violence Substance use | one year

CONTACTS AND LOCATIONS:
Overall Officials: Gregory L. Stuart, PhD, Principal Investigator — University of Tennessee-Knoxville & Butler Hospital; David Strong, PhD, Principal Investigator — Butler Hospital
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Stuart GL, McGeary J, Shorey RC, Knopik VS. Genetics moderate alcohol and intimate partner violence treatment outcomes in a randomized controlled trial of hazardous drinking men in batterer intervention programs: A preliminary investigation. J Consult Clin Psychol. 2016 Jul;84(7):592-8. doi: 10.1037/a0040219. Epub 2016 Mar 28. PMID 27018532